CLINICAL TRIAL: NCT06320197
Title: In Situ Simulation Training in Lifeguard Organisations: a Danish Retrospective Study From 2018-2023
Brief Title: In Situ Simulation Training in Lifeguard Organisations
Acronym: DROWN_INSITU
Status: Completed | Type: Observational
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Niklas Breindahl, Principal Investigator, Prehospital Center, Region Zealand
Other Study IDs: DROWN_INSITU
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Drowning; Drowning, Near; Drowning and Nonfatal Submersion; Drowning/Submersion; Drowning and Submersion While in Natural Water
Keywords: In situ simulation; Simulation; Drowning; Lifeguard; Lifesaver
MeSH Terms: conditions — Drowning; Near Drowning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Passed in situ assessment: This group passed their in situ assessment (summative assessment)
  Interventions: Other: In situ simulation assessment
- Failed in situ assessment: This group failed their in situ assessment (summative assessment)
  Interventions: Other: In situ simulation assessment

INTERVENTIONS:
Other: In situ simulation assessment — Unannounced in situ simulation assessment during working hours

SUMMARY:
This retrospective study will analyse a dataset consisting of 919 in situ simulation assessments collected between 2018 and 2023 in a Danish nationwide surf lifeguard organisation. The primary objective is to estimate the pass/fail ratio of in situ simulation assessments. The secondary objective is to analyse risk factors associated with a failed assessment. These results may guide future efforts to improve the Danish surf lifeguard training program.

DETAILED DESCRIPTION:
Background: Once weekly on all lifeguard-supervised beaches during the summer holiday period, a lifeguard instructor sneaks undetected into the primary surveillance zone between the flags and raises a hand to indicate a drowning scenario. This is called in situ simulation and is used to assess Danish surf lifeguards' rescue and medical skills. It is an unannounced test occurring during working hours, followed by feedback and training with the lifeguard instructors. Previous data indicate that approximately 1 in 5 lifeguards fail the in situ assessment. Analysing data from in situ simulation assessments may pinpoint areas for future improvement.

Objectives: The primary objective is to estimate the pass/fail ratio of in situ simulation assessments. The secondary objective is to analyse risk factors associated with a failed assessment. These results may guide future efforts to improve the Danish surf lifeguard training program.

Methods: This retrospective study will analyse a dataset consisting of 919 in situ simulation assessments collected between 2018 and 2023 in a Danish nationwide surf lifeguard organisation. Data on the local conditions (e.g., wave height, time of the day, and the number of beach visitors) and the in situ evaluation (pass/fail) were extracted directly from the predefined variables. Data on failure reasons were extracted through manual validation of the semi-structured free text fields by four independent observers. Any discrepancies were resolved by a senior member of the research group.

ELIGIBILITY:
Inclusion Criteria:

* All in situ assessments in the nationwide Danish lifeguard organisation from 2018 to 2023.

Exclusion Criteria:

* Blank entries
* Dublets

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants from this study are all trained in the nationwide Danish lifeguard organisation according to the International Life Saving Federations standards.
Sampling Method: Non-Probability Sample
Enrollment: 768 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pass/fail ratio of in situ simulation assessments | All in situ assessments from 2018-2023 will be included in this analysis.
  To estimate the pass/fail ratio of in situ simulation assessments.

SECONDARY OUTCOMES:
Risk factors associated with a failed assessment | All in situ assessments from 2018-2023 will be included in this analysis.
  To analyse risk factors associated with a failed assessment

CONTACTS AND LOCATIONS:
Overall Officials: Helle C Christensen, Ass. Prof., Study Director — Prehospital Center, Region Zealand
Locations (1):
- Prehospital Center, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will be available from the corresponding author upon reasonable request.